CLINICAL TRIAL: NCT05390866
Title: A Monocentric Randomised Controlled Trial to Investigate Changes in the Circulating Sphingolipidome Composition of Young and Healthy Individuals in Response to a Single Session of High-intensity Interval Training: the SphingoHIIT Study
Brief Title: Investigating the Circulating Sphingolipidome Response to a Single High-intensity Interval Training Session
Acronym: SphingoHIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Principal Investigator, Justin Carrard, Postdoctoral researcher, Principal investigator, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EKNZ 2022-00513
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Physiological Response of Sphingolipids to a Single HIIT Session
Keywords: Metabolomics; Lipidomics; High-intensity interval training; Ceramides; Sphingolipids; Cardiometabolic health

STUDY DESIGN:
Intervention Model Description: A prospective 2-arm, monocentric randomised controlled trial (a single HIIT session vs. no exercise intervention).
Who Masked: Participant, Investigator
Masking Description: Participants and investigators (except for the principal investigator) will also discover on the day of the HIIT intervention to which group they are allocated (HIIT vs. no exercise intervention). This information will be enclosed in a sealed envelope by the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIIT group (Experimental): The HIIT session will be conducted on a bicycle ergometer and consist of a 3-minute warm-up, followed by 4x4-minute intervals performed at 85-95% of the individually determined maximum heart rate, interspersed with 3-minute active recovery phases at a light effort). The HIIT session will be followed by a 2-minute cool-down phase.
  Interventions: Other: HIIT
- Control group (No Intervention): The control group will follow the same procedure except for the HIIT session, which will be replaced by a 30-minute physical rest in a sitting position. The participants will be allowed to read a book or work on their computer/phone.

INTERVENTIONS:
Other: HIIT — A single HIIT on a bicycle ergometer
  Arms: HIIT group

SUMMARY:
The purpose of this study is to examine the response of a comprehensive panel of circulating sphingolipids to a single high-intensity interval training (HIIT) session in healthy individuals in their twenties.

DETAILED DESCRIPTION:
Growing scientific evidence shows that specific sphingolipids, known as ceramides, predict cardiovascular risk beyond traditionally used biomarkers such as lipoproteins and triglycerides. Mechanistically, ceramides have been shown to promote foam cell formation, vascular inflammation, peripheral insulin resistance, and ultimately atherosclerosis. Currently, however, it remains unclear if and how physical activity, a simple, low-cost, and patient-empowering mean to optimise cardiometabolic health, can mitigate sphingolipid levels. The SphingoHIIT study aims to assess how certain circulating sphingolipid species respond to a single session of high-intensity interval training (HIIT). We hypothesise that circulating sphingolipid levels will be temporarily increased following a single HIIT session. This risk category A study will last 11 days and include 32 healthy participants aged between 20 and 29 years (50% of females). Participants will be randomly allocated either to the intervention group (n= 16) or the control group (n= 16). Blocked randomisation will be used to reduce bias and achieve balance in the allocation of participants to both groups, as commonly done when the sample size is small. Following an assessment of inclusion and exclusion criteria, a maximal cardiopulmonary exercise testing will be performed to determine peak oxygen uptake and peak heart rate. A washout period of five days will then be carried out before participants start to self-sample fasted dried blood spots to determine baseline levels of sphingolipids. After three days of sampling, participants will undergo a single HIIT session. Dried blood spots will be collected at five additional fixed time points (2min, 15min, 30min, 60min, and 24h) following the HIIT session. To minimise the dietary influence, participants will be asked to solely consume the provided individualised, pre-packaged meals starting one day before the first dried blood sampling.

Additionally, for the duration of the whole study, participants will wear a wrist accelerometer to track their physical activity. The SphingoHIIT study is expected to provide novel knowledge regarding the effect of an acute bout of physical exercise on sphingolipid levels. The results of this study will be published in a peer-reviewed journal and will be presented at scientific conferences.

ELIGIBILITY:
Inclusion Criteria:

* Female or male sex,
* Aged between 20 and 29 years old,
* Body Mass Index (BMI) between 18.5 and 24.9 kg/m2,
* Meeting the World Health Organization (WHO) guidelines on physical activity, i.e. at least 150-300 minutes of moderate-intensity aerobic physical activity per week as well as muscle-strengthening activities on 2 or more days per week,
* Clearance for physical activity according to the 2022 Physical Activity Readiness Questionnaire (PAR-Q+),
* Regular menstrual cycle,
* Informed consent as documented by signature.

Exclusion Criteria:

* Females with known pregnancy or breastfeeding,
* Females with known polycystic ovary syndrome (PCOS),
* Current exercise-limiting conditions of the lower limbs (e.g. tendinopathy, fractures or other musculoskeletal pathologies),
* Known acute or chronic diseases: e.g. any active infectious diseases, any past or current malignant tumours, any lung diseases (e.g. bronchial asthma), any cardiometabolic diseases (e.g. arterial hypertension, diabetes, dyslipidaemia), any gastrointestinal diseases (e.g. coeliac disease, Crohn's disease, ulcerative colitis), any psychological disorders (e.g. depression, if medically diagnosed, anorexia, bulimia), any endocrinological diseases (e.g. all types of diabetes mellitus, hyper- or hypothyroidism), any nephrological diseases, any neurological disorders,
* Current or past smoking, current or past psychoactive drug use (alcohol excluded here, see below),
* Excessive alcohol consumption in the past two weeks, defined as either binge drinking (consuming five or more drinks during a single occasion) or heavy drinking (consuming 15 or more drinks per week),
* Any current or regular medication use, including any kind of hormonal contraception,
* Diet: vegetarian, vegan, lactose-free and gluten-free, FODMAP-free (fermentable oligosaccharides, disaccharides, monosaccharides, and polyols),
* Inability to follow the procedures of the study, e.g. due to linguistic or cognitive problems,
* Concomitant involvement in another trial or participation in another trial in the last 4 weeks.

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Concentration of circulating Cer16:0, Cer18:0, Cer24:0 and Cer24:1 | 72 hours
  Quantifying the changes in serum level in the four sphingolipid species included in the ceramide-based scores (Cer16:0, Cer18:0, Cer24:0 and Cer24:1) following a single HIIT session.

SECONDARY OUTCOMES:
Concentration of the resting circulating sphingolipid species to be acquired | 72 hours
  Quantifying the changes in serum level in the resting sphingolipid species which will be acquired.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Prof, Study Chair — Department of Sport, Exercise and Health, University of Basel, Basel, Switzerland
Locations (1):
- Division of Sports and Exercise Medicine, Department of Sport, Exercise and Health, University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi RH, Tatum SM, Symons JD, Summers SA, Holland WL. Ceramides and other sphingolipids as drivers of cardiovascular disease. Nat Rev Cardiol. 2021 Oct;18(10):701-711. doi: 10.1038/s41569-021-00536-1. Epub 2021 Mar 26. PMID 33772258
- [Background] Laaksonen R, Ekroos K, Sysi-Aho M, Hilvo M, Vihervaara T, Kauhanen D, Suoniemi M, Hurme R, Marz W, Scharnagl H, Stojakovic T, Vlachopoulou E, Lokki ML, Nieminen MS, Klingenberg R, Matter CM, Hornemann T, Juni P, Rodondi N, Raber L, Windecker S, Gencer B, Pedersen ER, Tell GS, Nygard O, Mach F, Sinisalo J, Luscher TF. Plasma ceramides predict cardiovascular death in patients with stable coronary artery disease and acute coronary syndromes beyond LDL-cholesterol. Eur Heart J. 2016 Jul 1;37(25):1967-76. doi: 10.1093/eurheartj/ehw148. Epub 2016 Apr 28. PMID 27125947
- [Background] Tippetts TS, Holland WL, Summers SA. Cholesterol - the devil you know; ceramide - the devil you don't. Trends Pharmacol Sci. 2021 Dec;42(12):1082-1095. doi: 10.1016/j.tips.2021.10.001. Epub 2021 Nov 5. PMID 34750017
- [Background] Carrard J, Gallart-Ayala H, Weber N, Colledge F, Streese L, Hanssen H, Schmied C, Ivanisevic J, Schmidt-Trucksass A. How Ceramides Orchestrate Cardiometabolic Health-An Ode to Physically Active Living. Metabolites. 2021 Sep 30;11(10):675. doi: 10.3390/metabo11100675. PMID 34677390
- [Derived] Carrard J, Angst T, Weber N, Bienvenue J, Infanger D, Streese L, Hinrichs T, Croci I, Schmied C, Gallart-Ayala H, Hochsmann C, Koehler K, Hanssen H, Ivanisevic J, Schmidt-Trucksass A. Investigating the circulating sphingolipidome response to a single high-intensity interval training session within healthy females and males in their twenties (SphingoHIIT): Protocol for a randomised controlled trial. F1000Res. 2023 Aug 18;11:1565. doi: 10.12688/f1000research.128978.3. eCollection 2022. PMID 37533665